CLINICAL TRIAL: NCT06029595
Title: A 52-week, Randomised, Double Blind, Multicentre, 2-arm Parallel Group Trial Assessing Efficacy of CHF6001 (Total Daily Dose 3200μg) Dry Powder Inhaler (DPI) add-on to Maintenance Medium or High Dose of Inhaled Corticosteroids in Combination With Long-acting ß2-agonists in Subjects With Uncontrolled Asthma
Brief Title: Efficacy and Safety of Tanimilast in Asthmatics uNcontrolled on ICS-containinG backgrOund Maintenance Therapy
Acronym: TANGO
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Strategic decision by Sponsor; not due to safety reasons
Sponsor: Chiesi Farmaceutici S.p.A. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CLI-06001AA2-01; EUCT: 2022-502208-64-00 (Other: EU CTR)
Record Dates: First submitted 2023-08-31; First posted 2023-09-08 (Actual); Last update posted 2025-12-18 (Actual); Status verified 2025-03

CONDITIONS: Uncontrolled Asthma
Keywords: Asthma; PDE4 inhibitor; anti-inflammatory respiratory drug; Tanimilast
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Intervention Model Description: Randomised, double-blind, placebo-controlled, 2-arm parallel group study
Who Masked: Participant, Investigator
Masking Description: Double (Participant, Investigator)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CHF6001 - CHF6001 total daily dose 3200 μg; (Experimental)
  Interventions: Drug: Experimental: CHF6001 3200 μg
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo Comparator: CHF6001 Placebo

INTERVENTIONS:
Drug: Experimental: CHF6001 3200 μg — 800 μg/actuation - 2 inhalations of CHF6001 800 μg twice daily (BID) total daily dose 3200 μg
  Arms: CHF6001 - CHF6001 total daily dose 3200 μg;
Drug: Placebo Comparator: CHF6001 Placebo — 2 inhalations of CHF6001 matching placebo BID
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of CHF6001 (Tanimilast) as add-on to maintenance of inhaled corticosteroids in combination with Long-acting ß2-agonists in the target patient population. (TANGO)

ELIGIBILITY:
Inclusion Criteria:

1. Subject's written informed consent
2. Male or female subjects aged ≥18 and ≤75 years
3. A documented history of physician-diagnosed asthma for at least 1 year and with diagnosis before the age of 50 years
4. Stable asthma therapy: a stable maintenance treatment with medium to high dose of inhaled corticosteroids plus long acting β2 agonists for at least 3 months prior to screening
5. A prebronchodilator FEV1 ≤80% of the predicted normal value
6. Bronchodilator responsiveness after inhalation of salbutamol or equivalent
7. Evidence of poorly controlled or uncontrolled asthma as based on an ACQ-7 score ≥1.5
8. History of asthma exacerbations : at least 1 asthma exacerbation leading to hospitalisation or 2 or more asthma exacerbations within the last 12 months
9. A cooperative attitude and ability to use inhalers and to comply with study procedures

Exclusion Criteria:

1. e-Diary completion compliance <75% during run-in
2. History of near fatal asthma or of a past hospitalisation for asthma in intensive care unit
3. Recent exacerbation or respiratory tract infection within 4 weeks prior to screening visit or during the run-in period
4. Subjects using systemic corticosteroids medication in the 4 weeks or slow-release corticosteroids in the 12 weeks prior to randomisation
5. Asthma requiring use of biologics
6. Respiratory disorders other than asthma: subjects with known respiratory disorders other than asthma
7. Subjects with a history of lung volume resection
8. Current smokers, ex-smokers with a smoking history of ≥10 pack-years or current use of inhaled or oral cannabis products.
9. Subjects with cancer or history of cancer
10. Subjects with cardiovascular diseases
11. Subjects with any abnormal and clinically significant 12-lead ECG
12. Subjects with previous medical history, evidence of an uncontrolled intercurrent illness, or any clinically relevant abnormal findings in haematology, clinical chemistry, or urinalysis
13. Subjects with a diagnosis of depression, generalised anxiety disorder, suicidal ideation or behaviour
14. Patients mentally or legally incapacitated or patients accommodated in an establishment
15. Subjects with liver diseases
16. Drugs with hepatoxicity potential
17. Subjects with contra-indications to IMPs:
18. Subjects with history alcohol/drug abuse
19. Subjects with major surgery in the 3 months prior to screening visit or planned during the trial
20. Subjects treated with non-potassium sparing diuretics, nonselective β-blocking drugs, quinidine, quinidine like anti-arrhythmic, or any medication with a QTc prolongation potential or a history of QTc prolongation
21. Subjects treated with monoamine oxidase inhibitors (MAOIs) and tricyclic anti-depressants
22. Subjects receiving any therapy that could interfere with the study drugs
23. Participation in another investigational trial
24. Documented coronavirus disease 2019 (COVID-19) diagnosis within the last 2 weeks
25. Subjects having received a vaccination within 2 weeks prior to screening or during the run-in period.
26. For females only: pregnant or lactating women

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 517 (Actual)
Dates: Start 2023-11-26 (Actual); Primary Completion 2025-12-09 (Actual); Study Completion 2025-12-09 (Actual)

PRIMARY OUTCOMES:
Number of Asthma exacerbation over 52 weeks of treatment | Over 52 weeks
  Number of Asthma exacerbation over 52 weeks of treatment (Asthma exacerbations defined as severe event with worsening of asthma requiring at least 3 days of SCS use with or without emergency visit or hospitalization)

SECONDARY OUTCOMES:
Time to first asthma exacerbation; | Up to 52 weeks
  Asthma exacerbations defined as severe event with worsening of asthma requiring at least 3 days of SCS use with or without emergency visit or hospitalization
Number of asthma exacerbation and asthma worsening over 52 weeks of treatment | Up to 52 weeks
  Asthma exacerbations defined as severe event with worsening of asthma requiring at least 3 days of SCS use with or without emergency visit or hospitalization; Asthma worsening defined as moderate asthma exacerbation.
Time to first asthma exacerbation or asthma worsening | Up to 52 weeks
  Asthma exacerbations defined as severe event with worsening of asthma requiring at least 3 days of SCS use with or without emergency visit or hospitalization; Asthma worsening defined as moderate asthma exacerbation.
ACQ-7 responders | week 4, week 26 and week 52
  ACQ-7 responders at Week 4, Week 26 and Week 52 (i.e., subjects showing improvement from baseline in ACQ-7 score of ≥0.5 units);
Change from baseline in ACQ-7 and ACQ-6 | week 4, week 26 and week 52
  Change from baseline in ACQ-7 and ACQ-6 at Week 4, Week 26 and Week 52
Change from baseline in Mini-AQLQ | week 4, week 26 and week 52
  Change from baseline in Mini-AQLQ at Week 4, Week 26 and Week 52
Change from baseline in pre-dose FEV1 | week 4, week 26 and week 52
  Change from baseline in pre-dose FEV1 at Week 4, Week 26 and Week 52;
Change from baseline in pre-dose FVC | Week4, Week 52 and Week 26
  Change from baseline in pre-dose FVC at Week4, Week 52 and Week 26;
Change from baseline (run-in period) to each inter-visit period and to the entire treatment period in pre dose morning/evening PEF; | Up to 52 weeks
Change from baseline to each inter-visit period and to the entire treatment period in the average rescue medication use (number of puffs/day) and asthma symptoms score | Up to 52 weeks
Change from baseline to each inter-visit period and to the entire treatment period in the percentage of rescue medication-free days, asthma symptoms-free days and asthma control days. | Up to 52 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Johann Christian VIRCHOW, Prof, Principal Investigator — Universitätsmedizin Rostock
Locations (187):
- Argentina (32):
  - Site 032020 - Instituto Especialidades de la Salud Rosario - Clinica del Torax, Santa Fe, La
  - Site 032027- Centro de Medicina Respiratoria, Argentina
  - Site 032025 - Sala Mignaburu, Berazategui
  - Site 032004 - CARE - Centro de Alergia y Enfermedades Respiratorias, Buenos Aires
  - Site 032008 - Mautalen Salud e Investigacion, Buenos Aires
  - Site 032014 - Instituto de Investigaciones en Alergia y Enfermedades Respiratorias (INAER), Buenos Aires
  - Site 032021 - Centro De Investigaciones Medicas Mar Del Plata, Buenos Aires
  - Site 032024 -CEMLO- Consultorio Medico CEMLO LOBOS, Buenos Aires
  - Site 032029 - Hospital de Alta Complejidad del Bicentenario de Esteban Echeverría, Buenos Aires
  - Site 032030 - Instituto de Diagnostico e Investigaciones Metabolicas (IDIM), Buenos Aires
  - Site 032031 - Centro de Investigaciones Metabolicas (CINME) S.A., Buenos Aires
  - Site 032032 - Hospital Italiano de Buenos Aires (HIBA), Buenos Aires
  - Site 032003 -Fundacion Respirar (Centro Medico Dra. De Salvo) - Instituto Argentino de Investigaciones Clinicas (IAIC) S.R.L, Ciudad de Buenos Aires
  - Site 032026 - IAAER-Instituto de Asma, Alergia y Enfermedades Respiratorias, Corrientes
  - Site 032005 - National University of Cordoba - Rusculleda Foundation - Instituto DAMIC, Córdoba
  - Site 032010 - Centro Platense en Investigaciones Respiratorias - CEPIR, La Plata
  - Site 032013 - Centro de Investigacion Medico Lanus-CIMEL CHAHIN CHAHIN S.A, Lanús
  - Site 032006 -Institute Fundacion Enfisema - Instituto Ave Pulmo; Hospital Privado de Comunidad (HPC), Mar del Plata
  - Site 032002 -Consultorios Medicos Dr Isaac Scherbovsky - Fundacion Scherbovsky, Mendoza
  - Site 032009 - Centro Medico INSARES, Mendoza
  - Site 032023 - Respira Salud Clinica Integral, Mendoza
  - Site 032011 - Centro Privado de Medicina Respiratoria de Parana - CPMR, Paraná
  - Site 032007 - Instituto Especialidades de la Salud Rosario - Clinica del Torax, Rosario
  - Site 032016 - Instituto Medico de la Fundacion Estudios Clinicos, Rosario
  - Site 032019 - Servicio de Investigacion de Patologias Alergicas del Instituto ABC - Rosario, Rosario
  - Site 032001 - Instituto de Enfermedades Respiratorias e Investigacion Medica- IERIM, San Juan Bautista
  - Site 032015 - Fundacion de Estudios Clinicos de Consultorio Integrados Rosario, San Miguel de Tucumán
  - Site 032018 - Instituto de Investigaciones en Patologias Respiratorias, San Miguel de Tucumán
  - Site 032022 - Clinica Mayo de Urgencias Medicas Cruz Blanca SRL, San Miguel de Tucumán
  - Site 032012 - Instituto Del Buen Aire, Santa Fe
  - Site 032028 - Instituto De Investigaciones Clnicas De Rosario, Santa Fe
  - Site 032017 - Centro Medico de Enfermedades Respiratorias (CEMER), Vicente López
- Bulgaria (29):
  - Site 100012 - Medical Center Asklepii OOD, Dupnitsa
  - Site 100005 _MHAT Dr. Tota Venkova AD, Gabrovo
  - Site 100011 - Medical Center Pulmo-2018 EOOD, Haskovo
  - Site 100022 - MHAT Dr. Atanas Dafovski AD, Kardzhali
  - Site 100021 - MC Zdrave 1, Kozloduy
  - Site 100003 - """DCC 1 - Pernik"" EOOD", Pernik
  - Site 100010 - Medical Center FAMA, Plovdiv
  - Site 100017 - MHAT Sveti Panteleymon EOOD, Plovdiv
  - Site 100025 - Dr. Filip Shterev - Individual ambulatory practice for specialized medical care, Plovdiv
  - Site 100024 - Medical center Respiro, Razgrad
  - Site 100006 _ Ambulatory For Specialized Outpatient Medical Care - Individual Practice - Dr. Nikolay Evgeniev Ruse Ltd, Rousse
  - Site 100014 -SBALPFZ - Ruse EOOD, Rousse
  - Site 100029 - DCC 1 Sevlievo, Sevlievo
  - Site 100016 - MHAT Shumen AD, Shumen
  - Site 100004 - MHAT Dr. Ivan Seliminski AD, Sliven
  - Site 100028 - Smolyan Clinical Research Center, Smolyan
  - Site 100001- 5th MHAT - Sofia EAD, Sofia
  - Site 100002 _MHAT St. Ekaterina Dimitrovgrad, Sofia
  - Site 100008 _Diagnostic Consultative Center Convex Ltd, Sofia
  - Site 100013 - MHAT Lyulin EAD, Sofia
  - Site 100015 - Hospital for Pneumatic Physiatric Diseases - Sofia, Sofia
  - Site 100018 - Medical Center Excelsior Ltd, Sofia
  - Site 100019 - Aleksandrovska University Hospital, Sofia
  - Site 100020 -Medical Centre N. I. Pirogov EOOD, Sofia
  - Site 100023 - University First Multiprofile Hospital for Active treatment-Sofia EAD, Sofia
  - Site 100030 - Medical Center Hera EOOD, Sofia
  - Site 100009 - Medical Center Kissiovi, Varna
  - Site 100027 - Medical Center Research Expert, Varna
  - Site 100007 _SHATPPD Vratsa, Vratsa
- Czechia (10):
  - Site 203001 -MUDr. I. Cierna Peterova s.r.o., Brandýs nad Labem
  - Site 203008 - Fakultni nemocnice Brno, Brno
  - Site 203002 - MediTrial s.r.o., Jindřichův Hradec
  - Site 203009 - Alergologie Nemcova s.r.o, Lískovec
  - 203004 -Nemocnice Mesice, Měšice
  - Site 203006 - Nemocnice Znojmo, Ostrava
  - Site 203010 - DAWON Spol. s r.o. - Pneumologicka Ambulance, Prague
  - Site 203011 -Ordinace chorob plicnich s.r.o., Prague
  - Site 203003 - Plicni Stredisko Teplice, s.r.o., Teplice
  - Site 203005 - Ambulance Pneumologie a Ftizeologie, Varnsdorf
- Georgia (7):
  - Site 268001 - Chapidze Emergency Cardiology Center, Tbilisi
  - Site 268002 - JSC German Hospital, Tbilisi
  - Site 268003 - French Joint Hepatology Clinic Hepa, Tbilisi
  - Site 268004 - LTD Helsicore, Tbilisi
  - Site 268005 - LLC Medi Club Georgia, Tbilisi
  - Site 268006 - The Firsts University Clinic of Tbilisi State Medical University, Tbilisi
  - Site 268007 - TSMU & Ingorokva High Medical Technologies University Clinic, Tbilisi
- Germany (21):
  - Site 276004 - RCMS, Berlin
  - Site 276012 - Institut fuer Allergie- und Asthmaforschung Berlin, Berlin
  - Site 276013 - MECS Research, Berlin
  - Site 276010 - Office of Dr. Thomas Ginko, MD, Bonn
  - Site 276014 - MECS Cottbus GmbH, Cottbus
  - Site 276019 - Praxis Dr. Eckhardt, Delitzsch
  - Site 276007 - IKF Institut fuer klinische Forschung Frankfurt, Frankfurt am Main
  - Site 276008 - Office of Dr. med. Claus Keller MD, Frankfurt am Main
  - Site 276003 - ME Clinical Respiratory Research Hamburg, Hamburg
  - Site 276015 - Velocity Clinical Research Hamburg GmbH, Hamburg
  - Site 276002 - Pneumologicum im Suedstadtforum - Hannover, Hanover
  - Site 276009 - Velocity Clinical Research Leipzig GmbH, Leipzig
  - Site 276011 - POIS Sachsen GmbH, Leipzig
  - Site 276020 - BAG Prof. Gerhard Hoheisel/Dr. Andreas Bonitz Praxis für Pneumologie und Allergologie-Studienzentrum, Leipzig
  - Site 276006 - IKF Pneumologie Mainz, Helix Medical Excellence Center Mainz, Mainz
  - Site 276001 - Studienzentrum Muenchen-West; Gemeinschaftspraxis fuer Lungen- und Bronchialheilkunde Prof. Dr. med. Rainald Fischer und Dr. med. Michael Baborka, München
  - Site 276021 - Pneumologische Gemeinschaftspraxis Rheine, Rheine
  - Site 276022 - Universitaetsmedizin Rostock, Rostock
  - Site 276016 - Praxisgemeinschaft in Saalfeld - HNO, Saalfeld
  - Site 276018 - Siteworks Prufzentrum Schleswig-RespiRatio, Schleswig
  - Site 276005 - Lungenzentrum Ruhr - Praxis fuer Lungenheilkunde, Witten
- Hungary (5):
  - Site 348006 - Bajcsy-Zsilinszky Hospital, Budapest
  - Site 348003 - ClinTrial-Kenezy Hospital Institute of Clinical Pharmacology Infectology and Allergology, Debrecen
  - Site 348001 - Koch Robert Korhaz es Rendelointezet, Edelény
  - Site 348005 - Szalay Janos Rendelointezet, Hajdúnánás
  - Site 348004 - INFER-MED Kft. Da Vinci Maganklinika, Pécs
- Italy (6):
  - Site 380002 - AOU-S.Orsola-Malpighi - Universita degli Studi di Bologna, Bologna
  - Site 380003 - Azienda Ospedaliero Universitaria OO RR di Foggia, Foggia
  - Site 380001 - SC Pneumologia -Fondazione IRCCS Policlinico San Matteo, Pavia
  - Site 380006 - Azienda Ospedaliero Universitaria Pisana - Stabilimento Ospedaliero di Santa Chiara, Pisa
  - Site 380005 - Ospedale Fatebenefratelli Isola Tiberina Gemelli Isola, Roma
  - Site 380004 - Fondazione Salvatore Maugeri I.R.C.C.S. - Istituto Scientifico di Tradate, Tradate
- Latvia (7):
  - Site 428005 - Balvi and Gulbene hospital union, Balvi
  - Site 428008 - Dubultu Poliklinika, Jūrmala
  - Site 428001 - Pauls Stradins Clinical University Hospital, Riga
  - Site 428002 - Consilium Medicum SIA, Riga
  - Site 428003 - Latvian University Medical Postgraduate Institute, Riga
  - Site 428006 - RiGa 1st Hospital, Riga
  - Site 428007 - SIA RAKUS, Riga
- Lithuania (4):
  - Site 440002 - Hospital of Lithuanian University of Health Sciences Kauno klinikos, Kaunas
  - Site 440003 - LSMU Kauno ligoninė (Kaunas Hospital of the Lithuanian University of Health Sciences), Kaunas
  - Site 440006 - CD8 Klinika, Kaunas
  - Site 440001 - Viesoji Istaiga Antakalnio poliklinika, Vilnius
- Poland (23):
  - Site 616011 - Centrum Medycyny Oddechowej, Mroz Spolka Jawna, Bialystok
  - Site 616017 - NZOZ Przychodnia Vitamed, Bydgoszcz
  - Site 616024- Mital Site, Elblag
  - Site 616015 - Centrum Medyczne CLW-MED Aneta Cichomska i Joanna Luka-Wendrowska, Grudziądz
  - Site 616020 - Pro Familia Altera Sp. z o.o., Katowice
  - Site 616001 - Malopolskie Centrum Alergologii Sp z o.o, Krakow
  - Site 616018 - Prywatna Praktyka Lekarska Adam Śmiałowski - Intermed Ksawerów, Ksawerów
  - Site 616007 - ETG Lodz, Lodz
  - Site 616009 - Samodzielny Publiczny Zaklad Opieki Zdrowotnej Uniwersytecki Szpital Kliniczny Nr 1 im. Norberta Barlickiego Uniwersytetu Medycznego w Lodzi, Lodz
  - Site 616021 -IP Clinic Sp. z o.o., Lodz
  - Site 616008 - Centrum Alergologii Specjalistyczna Przychodnia Alergologiczna, Lublin
  - Site 616025 - MS Pneumed Janusz Milanowski, Katarzyna Szmygin-Milanowska Spolka Jawna, Lublin
  - Site 616022 - Makowskie Centrum Medyczne Hamernia Sp. z o.o., Maków Podhalański
  - Site 616013 - Ostrowieckie Centrum Medyczne Spolka Cywilna Anna Olech-Cudzik, Krzysztof Cudzik, Ostrowiec Świętokrzyski
  - Site 616006 - Centrum Alergologii Teresa Hofman Sp.z.o.o, Poznan
  - Site 616019 - Alergologia Plus, Poznan
  - Site 616023 - Specjalistyczna Przychodnia Lekarska Alergo-Med Sp. z o.o, Poznan
  - Site 616014 - Pawlukiewicz Malgorzata Prywatny Gabinet Lekarski, Rzeszów
  - Site 616004 - Centrum Medyczne Lucyna Andrazej Dymek - Strzelce Opolskie, Strzelce Opolskie
  - Site 616005 - Niepubliczny Zaklad Opieki Zdrowotnej (NZOZ) - Poradnia Chorob Pluc, Słupsk
  - Site 616003 - Lekarze Specjalisci - J. Malolepszy i Partnerzy, Wroclaw
  - Site 616012 - Centrum Badan Klinicznych Piotr Napora Lekarze Spolka Partnerska, Centrum Badan Klinicznych Osrodek Badan Wczesnej Fazy, Wroclaw
  - Site 616016 - Michal Bogacki Dobrostan, Wroclaw
- Romania (9):
  - Site 642005 - Angisan grup srl, Bragadiru
  - Site 642001 - Centrul Medical de Diagnostic si Tratament Neomed, Brasov
  - Site 642002 - Institute of Pneumology 'Marius Nasta', Bucharest
  - Site 642004 - Clinical Hospital Of Pneumology Leon Daniello, Cluj-Napoca
  - Site 642007 - ICRH Prof DR Octavian Fodor, Sectia Medicina Interna si Ambulator Alergologie, Cluj-Napoca
  - Site 642003 - Spitalul De Boli Infectioase Victor Babes, Craiova, Craiova
  - Site 642008 - SPITALUL CLINIC DE PNEUMOFTIZIOLOGIE IASI, Sectia Clinica I de Pneumologie, Iași
  - Site 642006 - Fundatia Cardioprevent, Timișoara
  - Site 642009 - Spitalul Clinic de Boli Infectioase si Pneumoftiziologie Dr. Victor Babes, Timișoara
- South Africa (16):
  - Site 710005 - Worthwhile Clinical Trials, Benoni
  - Site 710013 - Office of Dr. Agatha Cathrine Wilhase, MD, Boksburg
  - Site 710016 - Tsitsikamma Clinical Research Initiative, Cape Town
  - Site 710003 - Office of Dr. ZFA Vawda MD, Durban
  - Site 710004 - Synapta Clinical Research Center, Durban
  - Site 710012 - CRISMO Research Centre, Germiston
  - Site 710015 - University Of The Witwatersrand, Johannesburg
  - Site 710006 - Langeberg Medicross Medical Centre, Kraaifontein
  - Site 710002 - Lenmed- Ahmed Kathrada Private Hospital, Lenasia
  - Site 710007 - Ubuntu Clinical Research, Lenasia
  - Site 710001 - Emmed Research- Jakaranda Hospital, Pretoria
  - Site 710009 - Global Clinical Trials, Pretoria
  - Site 710011 - Busamed Paardevlei Hospital, Somerset West
  - Site 710014 - University Of Stellenbosch, Stellenbosch
  - Site 710010 - Limpopo Clinical Research Initiative, Thabazimbi
  - Site 710008 - Welkom Clinical Trial Centre, Welkom
- South Korea (10):
  - Site 410003 - Hallym University Sacred Heart Hospital, Anyang-si
  - Site 410012 - Chungbuk National University Hospital (CBNUH), Cheongju-si
  - Site 410004 - Jeonbuk National University Hospital, Jeonju
  - Site 410001 - Konkuk University Medical Center, Seoul
  - Site 410002 - The Catholic University of Korea, Seoul St. Marys Hospital, Seoul
  - Site 410005 - Korea University Guro Hospital, Seoul
  - Site 410006 - Asan Medical Center (AMC), Seoul
  - Site 410007 - Kangbuk Samsung Hospital, Seoul
  - Site 410008 - Severance Hospital, Yonsei University Health System, Seoul
  - Site 410009 - Ajou University Hospital, Suwon
- Spain (8):
  - Site 724005 - Clinica Mi Tres Torres Barcelona, Barcelona
  - Site 724008 - Hospital del SAS de Jerez de la Frontera, Jerez de la Frontera
  - Site 724007 - Hospital General Universitario Gregorio Maranon (HGUGM) - Instituto de Investigacion Sanitaria Gregorio Maranon (IiSGM), Madrid
  - Site 724002 - Servicio Andaluz de Salud Consejeria de Salud - Hospital Universitario Virgen de la Victoria, Málaga
  - Site 724004 - Hospital Universitario Marqués de Valdecilla, Santander
  - Site 724006 - Complejo Hospitalario Universitario De Santiago, Santiago de Compostela
  - Site 724003 - Hospital La Plana, Vila-real
  - Site 724001 - Hospital Universitario Miguel Servet, Zaragoza

IPD SHARING:
Plan to Share IPD: No